CLINICAL TRIAL: NCT03646656
Title: Heart Health Buddies: Peer Support to Decrease Cardiovascular Risk (CDA 13-263)
Brief Title: Heart Health Buddies: Peer Support to Decrease CVD Risk
Acronym: HHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 18-005
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular disease; social support
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- peer partner (Experimental): Veterans with at least one CVD risk factor who are interesting in increasing heart healthy behaviors through peer support
  Interventions: Behavioral: reciprocal peer support and non reciprocal coach support
- peer coach (Other): Veterans with at least one CVD risk factor who have made and sustained changes in diet or exercise in the past 3-6 months prior to enrollment. While the investigators will collect data on peer coach participants, their participation is primarily as part of intervention to examine the feasibility and benefit of adding peer coaching to a peer partner intervention.
  Interventions: Behavioral: reciprocal peer support and non reciprocal coach support

INTERVENTIONS:
Behavioral: reciprocal peer support and non reciprocal coach support — Peers and peer coaches provide mutual or one-way support to initiate and sustain behavioral improvements for cardiovascular health, with additional education from study staff.

SUMMARY:
This pilot study will use a hybrid reciprocal peer support and peer coach model to initiate and sustain heart-healthy behavioral changes in Veterans. Veterans who are at-risk for cardiovascular disease (CVD) will be enrolled in the study and paired with another Veteran to receive and provide social support around engaging in CVD risk reduction behaviors. Enrolled participants will be offered a series of 3 group sessions focused on CVD risk reduction, goal setting and action plan development. Between group sessions, peer partners will be asked to have weekly calls to discuss action plan challenges, explore options for problem solving, and provide encouragement and accountability for personal goals. Participants who do not engage in the group sessions or weekly phone calls, or who request additional help, will receive support from trained peer coaches. The goal of this pilot study is to evaluate the proof of concept for a hybrid reciprocal peer support (RPS) and peer coach intervention to improve heart healthy behaviors among Veterans at risk for CVD.

DETAILED DESCRIPTION:
A total of 24 Veterans enrolled at the Durham Veterans Affairs Medical Center will be screened and enrolled. Eligible Veterans are 35-64 years old, with at least one uncontrolled or poorly controlled risk factor for CVD. In addition, 3-6 veterans will be enrolled and trained as heart health peer coaches, with eligibility being 35-64 years old, with at least one documented CVD factor who have sustained improvement in physical activity or dietary change in the previous 3-6 months. All participants complete a baseline assessment, three structured group meetings, and a 12 week post-intervention assessment. At the first group, each participant creates a behavioral goal, and peer partners are paired with another Veteran based on behavioral goal and gender. They are expected to call their peer once a week to discuss progress or difficulty with their action plan and support each other with problem solving. Post enrollment and prior to the first group meeting, Peer coaches will have 3-5 hours of motivational and communication training with study staff focusing on skills such as active listening, non-directive support, eliciting change-talk, promoting incremental change, and patient confidentiality. Peer coaches will interact with peer buddies during a) group sessions, b) at a 6 week phone check-in, and c) on-going support if needed. Additional support will be initiated if there are no phone calls between pairs, there is a lack of participant engagement in calls to partner or attending group sessions, or upon request by the peer. There are two Aims of the current pilot study. Aim 1: examine the feasibility and acceptability of a 12-week hybrid peer coach-reciprocal peer support intervention. Feasibility will be evaluated by ease of recruitment, and enrollment and retention rates. Acceptability will be assessed by self-report of amount, frequency and modality of contacts, participation rates for group sessions, and through post-intervention qualitative interviews.

Aim 2: explore gender differences in feasibility/acceptability of the hybrid peer support model. Gender differences will be evaluated through qualitative comparison of participant reported experiences with intervention content as well as peer and group interactions by gender; and, quantitatively via exploration of differences in enrollment, retention, refusal reasons and frequency of peer contacts.

ELIGIBILITY:
Inclusion Criteria:

Peer partners and peer coaches:

* Enrolled in a Durham Veterans Administration Health Care System primary care clinic (including the women's health clinic)
* At risk for cardiovascular disease as defined by having at least one of the following:

  * Uncontrolled hypertension
  * history of obesity defined as (BMI >30)
  * uncontrolled non-insulin dependent diabetes mellitus
  * In addition, Peer coaches have made and sustained a behavioral change in past 3-6 months to improve heart health
* English as preferred language
* no significant hearing impairment
* lives approximately 30 minutes from the Durham Veterans affairs Medical Center
* agrees to attend regular visits per study protocol
* no contraindication to engage in at least moderate physical activity
* willing to use personal phone for peer and coach contacts

Exclusion Criteria:

* insulin-dependent diabetes
* serious mental illness defined as schizophrenia, bipolar disorder, dementia, active psychosis psychiatric hospitalization within the last 12 months or current high-risk suicide flag in their electronic medical record
* active substance use as documented in electronic or positive screening during telephone screening
* limited Life expectancy (<6 months) or severely ill defined as enrolled in hospice or actively undergoing chemotherapy or radiation therapy for cancer
* currently pregnant or planning to become pregnant in next 6 months

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Goldstein, MD MSPH, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be given personal feedback during the course of the study, such as during their baseline and 12 week assessments (weight, bp, and exercise scores), and via an activity monitor they will wear to monitor their daily activity. Participants will receive individual feedback, but as this is a feasibility study we do not intend to share study outcome results with participants.

RESULTS

PARTICIPANT FLOW:
Groups:
- Reciprocal Peer Partner: Veterans with at least one cardiovascular disease risk factor who are interested in increasing heart healthy behaviors through peer support receive phone-based weekly support from a reciprocal peer support partner and as needed help from a peer coach.
- Peer Coach: Veterans with at least one cardiovascular disease risk factor who have made and sustained changes in diet or exercise in the past 3-6 months prior to enrollment serve as peer coaches and provide supplemental one-way support to reciprocal peer partners as needed.
Period: Overall Study
Arm/Group | Reciprocal Peer Partner | Peer Coach
Started | 12 | 3
Attended 1st Group Session | 10 | 3
Completed | 9 | 3
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reciprocal Peer Partner | Peer Coach | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.42 (7.39) | 61.67 (2.08) | 55.87 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 3 | 0 | 3
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment
Description: Number of participants contacted, screened and enrolled in the pilot
Time Frame: 12 weeks
Population: Number of participants contacted for participation
Measure: Count of Participants; unit: Participants
Arm/Group | Reciprocal Peer Partner | Peer Coach
Number analyzed (Participants) | 50 | 10
Participants
  contacted but not screened | 25 | 7
  screened by not enrolled | 13 | 0
  consented | 12 | 3

2. Primary Outcome: Feasibility Retention
Description: Retention rates from consent to enrollment and from enrollment to completion of study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Reciprocal Peer Partner | Peer Coach
Number analyzed (Participants) | 12 | 3
Participants
  completed study | 9 | 3
  did not complete study | 3 | 0

3. Primary Outcome: Acceptability
Description: Acceptability of study based on successful peer buddy contacts per pair (not applicable to coaches) and participation in group sessions.
Time Frame: 12 weeks
Population: participants who attended at least 1 group session
Measure: Mean (Full Range); unit: group sessions attended per participant
Groups:
- Reciprocal Peer Partner: Veterans with at least one CVD risk factor who are interested in increasing heart healthy behaviors through peer support receive phone-based weekly support from a reciprocal peer support partner and as needed help from a peer coach.
- Peer Coach: Veterans with at least one CVD risk factor who have made and sustained changes in diet or exercise in the past 3-6 months prior to enrollment serve as peer coaches and provide supplemental one-way support to reciprocal peer partners as needed.
Arm/Group | Reciprocal Peer Partner | Peer Coach
Number analyzed (Participants) | 10 | 3
group sessions attended per participant | 2.1 [1 to 3] | 2 [1 to 3]

4. Primary Outcome: Acceptability - Weeks Contact With Peer Buddy
Description: Acceptability of study based on successful peer buddy contacts per pair (not applicable to coaches)
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Reciprocal Peer Partner
Number analyzed (Participants) | 10
weeks | 8.33 [6 to 10]

5. Secondary Outcome: Gender Differences - Retention
Description: Quantitative and qualitative gender differences in feasibility and acceptance will be evaluated through quantitative differences in enrollment, retention and frequency of peer contacts, and qualitative comparison of participant-reported experiences with intervention content, peer and group interactions by gender. Data are presented only for reciprocal peer partner group as this was pre-specified to compare outcomes between men and women in the reciprocal peer partner group. Thus, peer coaches are not described in this outcome.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Reciprocal Peer Partner - Female; Reciprocal Peer Partner - Male: Veterans with at least one cardiovascular disease risk factor who are interested in increasing heart healthy behaviors through peer support receive phone-based weekly support from a reciprocal peer support partner and as needed help from a peer coach.
Arm/Group | Reciprocal Peer Partner - Female | Reciprocal Peer Partner - Male
Number analyzed (Participants) | 6 | 6
Participants | 5 | 4

6. Secondary Outcome: Gender Differences-enrollment
Description: as for outcome 5
Time Frame: 12 weeks
Population: participants by gender contacted by invitation letter for study participation
Measure: Count of Participants; unit: Participants
Arm/Group | Reciprocal Peer Partner - Female | Reciprocal Peer Partner - Male
Number analyzed (Participants) | 29 | 21
Participants
  sent invitation letter by not reached by phone | 17 | 11
  reached by phone but not consented | 6 | 4
  consented | 6 | 6

7. Secondary Outcome: Gender Differences - Mean Contacts Per Buddy Pair
Description: Quantitative and qualitative gender differences in feasibility and acceptance will be evaluated through quantitative differences in enrollment, retention and frequency of peer contacts, and qualitative comparison of participant-reported experiences with intervention content, peer and group interactions by gender.
Time Frame: 12 weeks
Population: consented participants by gender
Measure: Mean (Full Range); unit: weeks
Arm/Group | Reciprocal Peer Partner - Female | Reciprocal Peer Partner - Male
Number analyzed (Participants) | 6 | 6
weeks | 9 [9 to 9] | 7.66 [6 to 10]

ADVERSE EVENTS:
Time Frame: time of consent to end of study participation, 12 weeks
Arm/Group | Reciprocal Peer Partner | Peer Coach
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 3/12 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reciprocal Peer Partner (N=12) | Peer Coach (N=3)
exacerbation of existing Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) — occurred after consent and before intervention initiation
passed gallstones (Eye disorders) | 1 (1) | 0 (0)
knee injury in snow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — surgery planned prior to consent
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03646656/Prot_000.pdf